CLINICAL TRIAL: NCT02187393
Title: Determining in Vitro Properties of Epithelial Cells From Individuals With Genetic Variants Associated With Idiopathic Pulmonary Fibrosis
Status: Withdrawn | Type: Observational
Why Stopped: Technical difficulties with the wet bench side of proposed studies.
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 13-3027; R01HL097163 (NIH)
Record Dates: First submitted 2014-03-13; First posted 2014-07-11 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Idiopathic Pulmonary Fibrosis; Healthy
Keywords: Epithelial cell function of cells from individuals with various genotypes
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * (3) tubes of blood
  * sample of cells from the nose
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators are trying to understand the role of specific genes in the function of airway surface cells. The investigators know that there are some common genetic markers that are associated with various lung diseases. However, most people with these genetic markers never develop any evidence of lung disease, so it is not understand how or if these markers play a role in disease. Investigators are asking healthy people to provide three (3) tubes of blood as well as a sample of cells from their nose. Investigators will use the blood sample to provide genetic information (specifically, presence or absence of alleles known to be associated with pulmonary fibrosis). Nose cells from individuals with the genetic markers that investigators are studying will be grown in the the lab to allow investigators to learn more about how the cells respond to various forms of environmental stress, such as exposure to cigarette smoke. The goal of this study is to understand how specific genes affect airway cell function.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years of age
2. Ability to provide informed consent
3. Patent bilateral nares

Exclusion Criteria:

1. Significant nasal or sinus disease precluding nasal brushing
2. A history of or ongoing epistaxis (nose-bleeding)
3. Acute upper respiratory illness
4. Ongoing treatment of respiratory or sinus illness with antibiotics
5. Pregnancy
6. Age less than 18 years
7. Infection with human immunodeficiency virus (HIV) or viral hepatitides (Hepatitis B, Hepatitis C)
8. Prior volunteer for the same study
9. Known diagnosis of cystic fibrosis or other ciliary disorder (example: primary ciliar dyskinesia)
10. Treatment with anticoagulants (examples: warfarin/coumadin, low molecular weight heparins, direct thrombin inhibitors such as dabigatran, anti-platelet agents such as P2Y12 inhibitors like clopidogrel and prasugrel, aspirin, ticagrelor, or factor Xa inhibitors such as rivaroxaban)
11. Known thrombocytopenia (example: immune thrombocytopenic purpura)
12. Ongoing chemotherapy
13. Known platelet dysfunction or bleeding diathesis/hemophilia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: normal healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
in vitro epithelial integrity measured by transepithelial electrical resistance (TEER), reported in ohms | 6 weeks
  The in vitro epithelial cell culture process will take approximately 4-6 weeks after the cells collected are thawed. (At the time of collection from study subjects, cells will be frozen until the time of thawing and culturing.) The in vitro epithelial process will take 6 weeks to differentiate epithelial monolayers at which time the tests of epithelial integrity can be performed. Study subjects themselves are not being followed.

SECONDARY OUTCOMES:
gene expression (DSP, MUC5B, genes associated with ER Stress), reported as "fold-change" or "CT mean" | 6 weeks
  Gene expression assays (designed by Taqman/Life Technologies) will be used to examine expression of genes that we believe are associated with pulmonary fibrosis -- specifically, various mucins (MUC5B, MUC5AC, DSP, and numerous genes associated with endoplasmic reticulum (ER) stress). This will be measured on epithelial monolayers derived in vitro from cells collected from study subjects. The differentiation of epithelial monolayers can take 3-6 weeks depending on the vagaries of the cell culture technique.

OTHER OUTCOMES:
Epithelial monolayer permeability (protein and cell permeability) | 6 weeks.
  Epithelial monolayer permeability as measured by dextran/protein and neutrophil traffic through monolayer in vitro. This will be measured on epithelial monolayers derived in vitro from cells collected from study subjects. The differentiation of epithelial monolayers can take 3-6 weeks depending on the vagaries of the cell culture technique.

CONTACTS AND LOCATIONS:
Overall Officials: David A Schwartz, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States